CLINICAL TRIAL: NCT01584310
Title: Validation of the STAMP Screening Tool For Pediatric Nutritional Risk To Be Used in the Ambulatory Setting.
Brief Title: Validation of the STAMP Screening Tool
Acronym: STAMP2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, raanan shamir, Chairman, Institute of Gastroenterology, Nutrition and Liver Diseases, Rabin Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MMC206-2011KCTIL
Record Dates: First submitted 2012-04-05; First posted 2012-04-24 (Estimated); Last update posted 2016-04-12 (Estimated); Status verified 2016-04

CONDITIONS: Malnutrition
Keywords: Nutritional assessment; children; malnutrition
MeSH Terms: conditions — Malnutrition | interventions — Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- STAMP using (Active Comparator): 100 boys and girls aged 1 to 6, attending Clalit Health Care Services Pediatric Centers, will undergo an assessment using the STAMP Tool; a questionnaire including 3 questions with a summary score, according to which the nutritional risk level shall be determined. These children shall also undergo a complete dietician assessment in order to examine the validity of the STAMP Tool.
  Interventions: Other: questionnaire STAMP and dietary
- No STAMP using (Placebo Comparator): 150 files shall be reviewed in the beginning of the research and after 6 months in order to estimate the change in medical staff's attention to nutritional status, by way of noting relevant diagnoses, reference to nutritional status- related tests and recording of anthropometric measurements.
  Interventions: Other: No STAMP using

INTERVENTIONS:
Other: questionnaire STAMP and dietary — Children will undergo a complete evaluation by an investigating dietician and assessment by the STAMP tool in order to determine the extent of the nutritional risk on a numerical scale. According to findings children will get the dietary recommendations.
  Arms: STAMP using
Other: No STAMP using — No intervention
  Arms: No STAMP using

SUMMARY:
Insufficient nutritional intake, with or without concomitant morbidity, leads to weight loss or insufficient weight gain, is related to an increase in morbidity and mortality and exposes the child to medical complications. In addition, obesity is also related to complications during hospitalization and complications in general, and therefore early identification of these children is extremely important. Studies show that malnutrition is frequent among children upon hospitalization, where the risk of pediatric nutritional deterioration increases, even in the presence of mild stress factors. This risk is frequent mainly among children that arrive at the hospital with an initial poor nutritional status. Improving the nutritional status as part of the standard of care already at the ambulatory setting might improve the prognosis of children when ill. In Israel, nutritional screening in not conducted among children since there is no proper validated screening tool. Study objectives: To test the accuracy of the STAMP Screening Tool for pediatric nutritional risk which is designed to be used by nurses, and to compare it to a complete nutritional assessment conducted by a dietician in Clalit Health Care Services clinics. In addition, the investigators wish to examine the effects of using a screening tool for nutritional risk on the medical staff's attention to the nutritional status; this is measured by the collection of nutritional status-related data and their recording in the patient file.

Methods: 100 boys and girls aged 1 to 6, attending Clalit Health Care Services Pediatric Centers, will undergo an assessment using the STAMP Tool; a questionnaire including 3 questions with a summary score, according to which the nutritional risk level shall be determined. These children shall also undergo a complete dietician assessment in order to examine the validity of the STAMP Tool. In addition, 150 files shall be reviewed in the beginning of the research and after 6 months in order to estimate the change in medical staff's attention to nutritional status, by way of noting relevant diagnoses, reference to nutritional status- related tests and recording of anthropometric measurements.

A statistical analysis to examine the validity of the STAMP Tool shall be carried out using the kappa test (K) (30). The effect of the STAMP Tool use shall be calculated using the chi square test.

ELIGIBILITY:
Inclusion Criteria:

1. children between 1 and 6 years old
2. children treated at the clinics participating in the study

Exclusion Criteria:

1. Lack of consent or lack of Hebrew proficiency
2. children that not receiving treatment in day hospitalization at any hospital

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2012-10; Primary Completion 2014-07 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Validity and reliability | 1 year
  The height / weight tables accepted in England, CDC (Centers for Disease Control) and WHO (World Health Organization) will be used in order to compare weight and height. The children will be divided into 3 nutritional risk groups: low, moderate and high according to the STAMP toll assessment and the results will be compared to the dietician's complete assessment.Nutritional assessment will include: demographic and medical data, daily nutritional intake, blood tests, anthropometric measurements, patient's ability to comply with the nutritional requirements related to his age etc.

SECONDARY OUTCOMES:
Validity and efficiency | one year
  Methods for testing the effect of STAMP tool use on the attitude of the medical staff to the nutritional status, measured by collection of data related to the nutritional status and recording them in the patient's file. In order to examine questionnaire acceptance by the medical staff, time period required to complete the questionnaire will be measured and in addition, the staff will be required to express their opinion regarding the speed and ease of using the questionnaire using the 4-point Likert scale. The staff will be asked about their subjective opinion about using the questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Raanan Shamir, Professor, Principal Investigator — Institute of Gastroenterology, Nutrition and Liver Diseases, Schneider Children's Medical Center of Israel